CLINICAL TRIAL: NCT00596609
Title: Effects of Intrathecal Morphine on Transcranial Electric Motor-Evoked Potentials in Patients Undergoing Posterior Spine Fusion
Brief Title: Intrathecal Morphine on Transcranial Electric Motor-Evoked Potentials
Acronym: EIM
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Paul Stricker, MD, Children's Anesthesiology Associates
Other Study IDs: 2007-4-5176
Record Dates: First submitted 2008-01-09; First posted 2008-01-17 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Trauma, Nervous System
Keywords: Injections, intrathecal; Transcranial; Spinal Fusion; Evoked Potentials, Motor
MeSH Terms: conditions — Trauma, Nervous System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Group 1 will be subjects who receive Intrathecal Morphine.
  Interventions: Drug: Intrathecal Morphine
- 2: Group 2 will be subjects who do not receive Intrathecal Morphine.

INTERVENTIONS:
Drug: Intrathecal Morphine — * In the IT morphine group, prior to IT morphine injection (within 15 minutes of the injection), the neurophysiologist will be asked to obtain a set of TceMEP recordings. The recordings collected at this time will be labeled "Baseline." These will serve as controls for subsequent recording comparisons.
  * In the IT morphine group, the time of IT morphine injection will be recorded, as well as the dose. A timer will be started. The neurophysiologist will then be asked to collect four additional sets of TceMEP recordings, at 5, 10, 20, and 30 minutes after morphine injection.
  Groups: 1

SUMMARY:
Patients undergoing posterior spinal fusion (PSF) procedures for scoliosis are at risk for iatrogenic neurologic injury of the spinal cord and/or spinal nerve roots during surgical correction of the abnormal spinal curvature. The degree of neurologic injury can range from minor sensory deficits to complete paraplegia. Surgeons at CHOP utilize neurophysiologists to identify impending neurologic injury. These consultants monitor spinal cord pathways by recording and analyzing evoked potentials during the operation. Evoked potentials are low voltage electrical signals generated in response to transcranial or transcutaneous electrical stimulation of motor and sensory neural pathways.

Some patients undergoing PSF receive an injection of morphine into the cerebrospinal fluid during the operation. This intrathecal (IT) morphine has potent analgesic effects. While most commonly used anesthetic agents have well-characterized effects on evoked potentials, little data exists on the effects of IT morphine on transcranial electric motor-evoked potentials (TceMEPs).

This is a prospective observational study to characterize the effects of IT morphine on TceMEPs.

DETAILED DESCRIPTION:
Posterior spinal fusion surgery (PSF) is associated with significant postoperative pain. Numerous postoperative pain management strategies have been employed for patients undergoing these procedures, including continuous narcotic infusions, intravenous patient-controlled opioid analgesia, epidural analgesia, intrathecally administered narcotics, and combinations of these regimens. Most patients at CHOP have their pain managed with intravenous patient-controlled opioid analgesia alone or in combination with a single dose of intra-operatively administered intrathecal (IT) morphine.

Patients undergoing spinal fusion procedures are also at risk for perioperative neurologic injury. Surgeons at CHOP and other institutions routinely utilize neurophysiologists to evaluate at-risk neural pathways to identify impending spinal cord and spinal nerve root injury. These consultants monitor motor and sensory pathways by recording and analyzing evoked potentials and electromyography during the operation. Evoked potentials are low voltage electrical signals generated in response to transcranial or transcutaneous electrical stimulation of motor and sensory nerves.

At CHOP, IT morphine is injected by the surgeon after the scoliotic curvature has been corrected and spinal instrumentation is complete. This injection therefore occurs after the critical period for neurophysiologic monitoring and risk of spinal cord injury. It is injected after the neurophysiologist has given a reassuring assessment of neural integrity. This injection is given to patients who have spinal fusions extending below the second lumbar vertebral body. Injections are limited to this group of patients because the appropriate intervertebral spaces for intrathecal injection are not exposed in procedures that do not extend below this level.

Most commonly used anesthetic agents have well-characterized effects on evoked potentials. The effects of IT morphine on sensory-evoked potentials have been studied. However, little data exist on its effects on transcranial electric motor-evoked potentials. This study aims to characterize these effects; we hypothesize that intrathecal morphine has no effect on transcranial electric motor-evoked potentials in the doses used at our institution.

ELIGIBILITY:
Inclusion Criteria:

Intrathecal Morphine Group:

1. All patients with idiopathic scoliosis aged 11 through and including 18 who present to CHOP for posterior spinal fusion will be eligible
2. Patients with procedures anticipated to extend to or below the second lumbar vertebral level
3. Only patients given intrathecal morphine after curve correction and instrumentation will be studied

Control Group:

1. All patients with idiopathic scoliosis aged 11 through and including 18 who present to CHOP for posterior spinal fusion will be eligible
2. Patients with procedures not anticipated to extend to or below the second lumbar vertebral level
3. Patients who do not receive IT morphine injection as part of their routine anesthetic care

Exclusion Criteria:

Intrathecal Morphine Group:

1. Patients who receive inhaled anesthetic agents before or during the 30 minutes following IT morphine injection
2. Patients who receive neuromuscular blocking drugs within an hour before or during the 30 minutes following IT morphine injection.
3. Patients who develop significant changes in TceMEPs prior to intrathecal morphine injection
4. Patients with intraoperative hemodynamic instability which requires continuous vasoactive drug infusion (e.g., dopamine)
5. Patients with neuromuscular, congenital, or other non-idiopathic scoliosis
6. Pregnant or lactating females

Control Group:

1. Patients who receive inhaled anesthetic agents before or during the 30 minutes following IT morphine injection
2. Patients who receive neuromuscular blocking drugs within an hour before or during the 30 minutes following IT morphine injection.
3. Patients who develop significant changes in TceMEPs prior to the study interval
4. Patients with intraoperative hemodynamic instability which requires continuous vasoactive drug infusion (e.g., dopamine)
5. Patients with neuromuscular, congenital, or other non-idiopathic scoliosis
6. Pregnant or lactating females

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ages 11-18 with idiopathic scoliosis who are scheduled to have a posterior spinal fusion.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To quantitatively evaluate the effects of IT morphine on TceMEP amplitude and latency in patients undergoing PSF who have IT morphine injected after instrumentation | 30 minute period - Group 1 - after IT morphine injection or during skin closure for Group 2.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stricker, MD, Principal Investigator — Children's Anesthesiology Associates, Ltd.
Locations (1):
- The Children's Hospital of Philadephia, Philadelphia, Pennsylvania, United States